CLINICAL TRIAL: NCT03562429
Title: The Efficacy of TGF for Treating Osteoarthritis of the Knee: A Randomized Double-blind Controlled Trial
Brief Title: The Efficacy of TGF for Treating Osteoarthritis of the Knee
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Hen-Hong Chang, Professor, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMUH107-REC2-044
Record Dates: First submitted 2018-05-10; First posted 2018-06-19 (Actual); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: 180 subjects are divided into treatment group and control group (placebo).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TGF group (study group) (Experimental): Use TGF to treat osteoarthritis of the knee, 5g/time, 3 times a day, for 12 weeks.
  Interventions: Drug: TGF
- TGFP group (placebo group) (Placebo Comparator): Use TGFP to treat osteoarthritis of the knee, 5g/time, 3 times a day, for 12 weeks.
  Interventions: Drug: TGFP

INTERVENTIONS:
Drug: TGF — TGF is a powder formulation of Hu-Qian Wan (HQW). HQW is composited of 10 herbs, Chinemys reevesii (Gray), Phellodendron chinense Schneid., Achyranthes bidentata Blume, Anemarrhena asphodeloides Bunge, Rehmannia glutinosa Libosch., Paeonia lactiflora Pall., Cynomorium songaricum Rupr., Angelica sinensis (Oliv.) Diels, Citrus reticulata Blanco and Zingiber officinale Rosc..
  Other Names: Hu-Qian Wan
  Arms: TGF group (study group)
Drug: TGFP — TGFP is 1/20 concentration of Hu-Qian Wan (HQW). HQW is composited of 10 herbs, Chinemys reevesii (Gray), Phellodendron chinense Schneid., Achyranthes bidentata Blume, Anemarrhena asphodeloides Bunge, Rehmannia glutinosa Libosch., Paeonia lactiflora Pall., Cynomorium songaricum Rupr., Angelica sinensis (Oliv.) Diels, Citrus reticulata Blanco and Zingiber officinale Rosc..
  Other Names: the placebo of Hu-Qian Wan
  Arms: TGFP group (placebo group)

SUMMARY:
This study is to evaluate the efficacy of herbal formula TGF treating knee joint osteoarthritis(KOA) and its biochemical mechanism. The study design is a parallel randomized, placebo-controlled, double-blind clinical trial includes 180 patients with KOA. The patients are random allocated into study group(taking TGF) and control group(taking 1/20 TGF). After the 12 weeks treatment course, another 4 weeks is to follow-up the condition without medication. Assessments will be performed before and after treatment and the end of follow-up period.

The inclusion criteria are (1) age between 50~75 years old, (2) diagnosis of osteoarthritis: The Clinical/Radiographic classification criteria of American College of Rheumatology, American College of Rheumatology, (3) chronic knee pain over 3 months. The exclusion criteria are (1) the past history with systemic joint disease, such as autoimmune disease, (2) the patient with history of knee surgery or waiting for the total knee replacement, (3) any disease that affect the function of lower extremities, such as trauma, tumor or compensation of abnormal posture, (4) the condition that cannot participate this study, (5) the subjects non-compliance with the protocol.

The Assessments including primarily the WOMAC (VAS version, 3.1), VAS and the used dosage of Celebrex before and after treatment. The secondary assessments are (1) X ray, (2) Constitution in Chinese Medicine Questionnaire, (3) Short From-36, (4) erythrocyte sedimentation rate and C reactive protein, (5) Biomarkers: C-telopeptide of type II collagen, cartilage oligomeric matrix protein, Osteocalcin, Leptin, Interleukin-1, Interleukin-6, matrix metalloproteinase-3, matrix metalloproteinase-13, ADAMTS-4, transglutaminase-2, and (6) metabolomics.

DETAILED DESCRIPTION:
Introduction Knee osteoarthritis is a common disease of joint degeneration. Chronic inflammation is the major cause of this disease. One-third of the people over 65 years of age have Knee OA and the prevalence in women is more than in men. One-third of the people over 65 years of age have Knee OA and the prevalence in women is more than in men. The risk factors include age, weight, genetic factor, sex, bone density, and the past history of trauma or work. The more important risk factors are age and weight. These multiple factors make the change of knee joint, like chronic inflammation, joint remodeling and loss of function that make the change of joint homeostasis.

The diagnosis criteria of knee OA is based on two groups. In 1957, Kellgren and Lawrence established the criteria of radiological assessment and in 1986, Altman's group created the criteria of classification of idiopathic knee OA. In the beginning, only four pictures presented the four grade of knee OA without description. In 1963, Lawrence wrote the original description. Altman and his team used clinical signs combined with laboratory or radiography to established the diagnosis criteria. Now, the most used method is clinical and radiographic examination. In the clinical part, the patient should have knee pain with at least one of three items: age over than 50 years, the time of morning stiffness is less than 30 minutes or crepitus. In the radiography, the patient's X ray should show the definite osteophytes. The sensitivity can reach 91 percent and the specificity can reach 86 percent.

Knee joint is a diarthrodial joint. Two adjacent bones are covered by a layer of specialized articular cartilage and are encased in a connective tissue capsule lined by a synovial membrane, consisting of a thin cell layer of macrophages and fibroblasts. The main structural elements of knee include the articular cartilage (with chondrocytes), tidemark (separating the calcified and articular cartilage), calcified cartilage, and subchondral cortical and trabecular bone. The advanced osteoarthritic changes characterized by fissuring and fragmentation of the articular cartilage, chondrocyte proliferation and hypertrophy, duplication and advancement of the tidemark, expansion of the zone of calcified cartilage, thickening of the subchondral cortical plate and vascular invasion of the bone and calcified cartilage.

The signaling of cytokine is an important part of progression of knee OA. The initial is inflammation, maybe from cartilage or synovium. Then the hypertrophic chondrocyte and the macrophage of synovium will secret IL-1, 4, 13, TNF-α,β, MMP1,13 and ADAMTS 4, 5. The major function of MMP and ADAMTS is to degrade the articular cartilage.

The treatment of knee OA by OARSI (Osteoarthritis Research Society International) has one core treatment and four recommend treatment by different OA types. The core treatment includes strength training and exercise, weight management and education. The recommend treatment includes NSAIDs by oral or topical, acetaminophen, corticosteroid and duloxetine.

Drug treatments are mostly related to relief of symptoms and there is no disease-modifying OA drug approved by the agencies. And the side effects of NSAIDs. In the GI tract, the patient may have nausea, dyspepsia, heartburn and diaphragm disease. In the kidney, there are acute or chronic renal failure with dose/duration-dependent effect. But the side effect of topical NSAIDs is less than oral NSAIDs in the GI tract.

With regard to the description of Knee OA in ancient China, the symptoms of knee OA have been recorded in the Huangdi Neijing 2000 years ago. APLD is an old formula since Tang dynasty about 1200 years ago. In the rat models, it is effective in terms of the proliferation of cartilage chondrocytes and the damaged knee joint tissue repairing.

Based on the evidence, there are 10 clinical trials to study the effect of TCM in the KOA since 2004. The effect of TCM in improving symptoms of knee OA is similar with it of NSAIDs and better than glucosamine sulfate. The major effect is pain relief and the special effect is improving muscle strength that NSAIDs cannot do. The results are usually the improvement of symptoms but there are no the bio- mechanisms of TCM. 2016, Chen et al. published a meta-analysis about TCM and knee OA. There are 23 studies that include 2362 subjects. 18 of the studies showed significantly improved VAS pain scores, six of the studies showed significantly improved WOMAC pain subscale scores, and 16 of the trials showed significantly improved total effectiveness rates. But in the quality of these studies, only "incomplete outcome data" can reach "Low risk of bias" and other items get "high risk of bias" or "unclear risk of bias".

The researches of animal models and cell lines presented that the herbs have the ability of analgesic effect, anti-inflammation, the regulation of cell cycle (apoptosis), anti- oxidation and anti-degradation. Like ginseng, ginseng Rb1 decreases the inflammation by decreasing IL-1b, decreases degradation of cartilage by decreasing MMP-1, 13 and increasing collagen type II and improves cell differentiation process by Notch signaling. Resveratrol from cranberries and grapes has effects of anti-inflammation by decreasing IL-1b, TNF-a, COX-2 and NF-kB and regulate the homeostasis of cartilage by increasing collagen II and decreasing MMP-13. Pharmacological actions of herbs include decrease of substance P, inhibition of vascular endothelial growth factor, promotion of chondrocyte proliferation and vasodilation. These actions are different from the effects of NSAIDs.

Although the design and methodology of the 10 studies are gradually improving, the quality of these studies is still not enough. But the potential of Chinese medicine is still huge. According to the statement above, researchers should focus on the whole knee joint including skin, fat, vessel, nerve, muscle, synovium, ligament, bone and cartilage. TCM formula usually composited of various herbs which may affect different tissues of knee joint and play a synergic effect. The DMOADs of Chinese medicine is a novel prospect.

Methods and Materials This study is to evaluate the efficacy of herbal formula TGF treating knee joint osteoarthritis(KOA) and its biochemical mechanism. The study design is a parallel randomized, placebo-controlled, double-blind clinical trial includes 180 patients with KOA. The patients are random allocated into study group(TGF) and control group(TGFP). After the 12 weeks treatment course, another 4 weeks is to follow-up the condition without medication. Assessments will be performed before and after treatment and the end of follow-up period.

The inclusion criteria are (1) age between 50~75 years old, (2) diagnosis of osteoarthritis: The Clinical/Radiographic classification criteria of American College of Rheumatology, American College of Rheumatology, (3) chronic knee pain over 3 months. The exclusion criteria are (1) the past history with systemic joint disease, such as autoimmune disease, (2) the patient with history of knee surgery or waiting for the total knee replacement, (3) any disease that affect the function of lower extremities, such as trauma, tumor or compensation of abnormal posture, (4) the condition that cannot participate this study, (5) the subjects non-compliance with the protocol.

The primary outcomes are the WOMAC (VAS version, 3.1), VAS for pain and the used dosage of Celebrex before and after treatment. The WOMAC is the VAS version, 3.1 and divided into three sub-scales -- pain, stiffness and function. Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing. Stiffness (2 items): after first waking and later in the day. Physical Function (17 items): stair use, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy household duties, light household duties. Each item has 0-100 mm to evaluate the status and the higher values represent a worse outcome. These three sub-scales were summed to a total score (0-2400 mm). Visual analogue scale for pain is to evaluate the status of knee pain when check point. Using 0-100 mm scale is to evaluate knee pain by visual analogue scale. "0" is no pain and "100" is the worst pain that subjects had experienced before. The subject gives the value under the moment of check point. The used dosage of Celebrex is another method to evaluate the situation of pain in a period.

The secondary outcomes are X ray, Constitution in Chinese Medicine Questionnaire (CCMQ), WHOQOL-BREF, erythrocyte sedimentation rate, high-sensitive C reactive protein, Biomarkers (C-telopeptide of type II collagen, cartilage oligomeric matrix protein, Osteocalcin, Leptin, Interleukin-1, Interleukin-6, matrix metalloproteinase-3, matrix metalloproteinase-13, ADAMTS-4, transglutaminase-2), metabolomics and mitochondrial function. The X ray are taken in the baseline, the 12th weeks and the 16th weeks to evaluate the change after treatment. The Constitution in Chinese Medicine Questionnaire (CCMQ) is to evaluate the constitution. This scale (Constitution in Chinese Medicine Questionnaire) includes nine constitutions and each constitution has 6-8 items that used 1-5 points to evaluate the degree. "1" means "better" and "5" means "worse". The transformed points is equal to [(original points - the number of items)/(the number of items*4) ]*100. The WHOQOL-BREF is to evaluate the quality of life. This scale is "World Health Organization Quality of Life - BREF". It contains 4 domains (Physical health, Psychological, Social relationships and Environment) and 26 items ("1" means "worse" and "5" means "better"). This scale used the following steps to calculate the transformed points: 1.Check all 26 items from assessment have a range of 1-5, 2.Reverse 3 negatively phrased items, 3.Compute domain scores, 4. Delete cases with >20% missing data, 5.Check domain scores. Erythrocyte Sedimentation Rate (ESR) actually measures the rate of fall (sedimentation) of erythrocytes (red blood cells) in a sample of blood that has been placed into a tube. Results are reported as the millimeters of clear fluid (plasma) that are present at the top portion of the tube after one hour. The higher value means more inflammation. High-sensitivity C-reactive Protein is a protein that increases in the blood with inflammation and infection as well as following a heart attack, surgery, or trauma. Thus, it is one of several proteins that are often referred to as acute phase reactants. The high-sensitivity CRP test measures low levels of CRP in the blood to identify low levels of inflammation that are associated with risk of developing cardiovascular disease (CVD). The concentration of C-Telopeptide of Type II Collagen (CTX-II), Cartilage Oligomeric Matrix Protein (COMP), Osteocalcin, Leptin, interleukin-1 (IL-1), interleukin-6 (IL-6), matrix metalloproteinase-3 (MMP-3), matrix metalloproteinase-13 (MMP-13), a disintegrin and metalloproteinase with thrombospondin motifs-4 (ADAMTS-4) and Transglutaminase 2 (TG-2) are evaluated by ELISA kit. About the metabolite of the drugs, this measurement used LC-MS to get the molecular weight of Chinese herbal metabolites form blood, urine and synovial fluid. This method can help to identify the active substance from the formula (TGF). But now, the exactly active substance is unclear. About mitochondrial function, this study will focus on mtDNA copy number, the expression of mRNA in PGC-1α, NRF1 and mtTFA by quantitative polymerase chain reaction, the expression of protein in PGC-1α, NRF1 and mtTFA by Western blotting and anti-oxidant capacity by OxiSelectTM Trolox Equivalent Antioxidant Capacity (TEAC) Assay Kit (ABTS).

ELIGIBILITY:
Inclusion Criteria:

1. age between 50~75 years old
2. diagnosis of osteoarthritis: The Clinical/Radiographic classification criteria of American College of Rheumatology, ACR
3. chronic knee pain over 3 months.

Exclusion Criteria:

1. the past history with systemic joint disease, such as autoimmune disease
2. the patient with history of knee surgery or waiting for the total knee replacement
3. any disease that affect the function of lower extremities, such as trauma, tumor or compensation of abnormal posture
4. the condition that cannot participate this study
5. the subjects non-compliance with the protocol

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Western Ontario & McMaster Universities Osteoarthritis Index | Change from Baseline WOMAC VAS version 3.1 at 3 months
  This scale is the VAS version, 3.1 and divided into three sub-scales -- pain, stiffness and function. Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing. Stiffness (2 items): after first waking and later in the day. Physical Function (17 items): stair use, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy household duties, light household duties. Each item has 0-100 mm to evaluate the status and the higher values represent a worse outcome. These three sub-scales were summed to a total score (0-2400 mm).
Visual Analogue Scale for pain | Change from Baseline Visual Analogue Scale for pain at 3 months
  To evaluate the status of knee pain when check point. Using 0-100 mm scale is to evaluate knee pain by visual analogue scale. "0" is no pain and "100" is the worst pain that subjects had experienced before. The subject gives the value under the moment of check point.
the used dosage of Celebrex | Change from Baseline the used dosage of Celebrex at 3 months
  To evaluate the dosage of Celebrex when check point
Western Ontario & McMaster Universities Osteoarthritis Index | Change from Baseline WOMAC VAS version 3.1 at 4 months
  This scale is the VAS version, 3.1 and divided into three sub-scales -- pain, stiffness and function. Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing. Stiffness (2 items): after first waking and later in the day. Physical Function (17 items): stair use, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy household duties, light household duties. Each item has 0-100 mm to evaluate the status and the higher values represent a worse outcome. These three sub-scales were summed to a total score (0-2400 mm).
Visual Analogue Scale for pain | Change from Baseline Visual Analogue Scale for pain at 4 months
  To evaluate the status of knee pain when check point. Using 0-100 mm scale is to evaluate knee pain by visual analogue scale. "0" is no pain and "100" is the worst pain that subjects had experienced before. The subject gives the value under the moment of check point.
the used dosage of Celebrex | Change from Baseline the used dosage of Celebrex at 4 months
  To evaluate the dosage of Celebrex when check point

SECONDARY OUTCOMES:
X ray | Change from Baseline X ray at 3 months
  knee joint that associated with this study
X ray | Change from Baseline X ray at 4 months
  knee joint that associated with this study
Constitution in Chinese Medicine Questionnaire, CCMQ | Change from Baseline CCMQ at 3 months
  For evaluating the constitution. This scale (Constitution in Chinese Medicine Questionnaire) includes nine constitutions and each constitution has 6-8 items that used 1-5 points to evaluate the degree. "1" means "better" and "5" means "worse". The transformed points is equal to [(original points - the number of items)/(the number of itmes*4) ]*100.
Constitution in Chinese Medicine Questionnaire, CCMQ | Change from Baseline CCMQ at 4 months
  For evaluating the constitution. This scale (Constitution in Chinese Medicine Questionnaire) includes nine constitutions and each constitution has 6-8 items that used 1-5 points to evaluate the degree. "1" means "better" and "5" means "worse". The transformed points is equal to [(original points - the number of items)/(the number of itmes*4) ]*100.
WHOQOL-BREF | Change from Baseline WHOQOL at 3 months
  For evaluating the quality of life. This scale is "World Health Organization Quality of Life - BREF". It contains 4 domains (Physical health, Psychological, Social relationships and Environment) and 26 items ("1" means "worse" and "5" means "better"). This scale used the following steps to calculate the transformed points: 1.Check all 26 items from assessment have a range of 1-5, 2.Reverse 3 negatively phrased items, 3.Compute domain scores, 4. Delete cases with >20% missing data, 5.Check domain scores.
WHOQOL | Change from Baseline WHOQOL at 4 months
  For evaluating the quality of life. This scale is "World Health Organization Quality of Life - BREF". It contains 4 domains (Physical health, Psychological, Social relationships and Environment) and 26 items ("1" means "worse" and "5" means "better"). This scale used the following steps to calculate the transformed points: 1.Check all 26 items from assessment have a range of 1-5, 2.Reverse 3 negatively phrased items, 3.Compute domain scores, 4. Delete cases with >20% missing data, 5.Check domain scores.
ESR | Change from Baseline ESR at 3 months
  For evaluating the status of inflammation. Erythrocyte Sedimentation Rate (ESR) actually measures the rate of fall (sedimentation) of erythrocytes (red blood cells) in a sample of blood that has been placed into a tube. Results are reported as the millimeters of clear fluid (plasma) that are present at the top portion of the tube after one hour. The higher value means more inflammation.
ESR | Change from Baseline ESR at 4 months
  For evaluating the status of inflammation. Erythrocyte Sedimentation Rate (ESR) actually measures the rate of fall (sedimentation) of erythrocytes (red blood cells) in a sample of blood that has been placed into a tube. Results are reported as the millimeters of clear fluid (plasma) that are present at the top portion of the tube after one hour. The higher value means more inflammation.
CTX-II | Change from Baseline CTX-II at 3 months
  This study uses ELISA kit to measure the concentraion (pg/ml) of C-Telopeptide of Type II Collagen (CTX-II) .
CTX-II | Change from Baseline biomarkers at 4 months
  This study uses ELISA kit to measure the concentraion (pg/ml) of C-Telopeptide of Type II Collagen (CTX-II) .
COMP | Change from Baseline biomarkers at 3 months
  This study uses ELISA kit to measure the concentraion (ng/ml) of Cartilage Oligomeric Matrix Protein (COMP) .
COMP | Change from Baseline biomarkers at 4 months
  This study uses ELISA kit to measure the concentraion (ng/ml) of Cartilage Oligomeric Matrix Protein (COMP) .
Osteocalcin | Change from Baseline biomarkers at 3 months
  This study uses ELISA kit to measure the concentraion (ng/ml) of Osteocalcin .
Osteocalcin | Change from Baseline biomarkers at 4 months
  This study uses ELISA kit to measure the concentraion (ng/ml) of Osteocalcin .
Leptin | Change from Baseline biomarkers at 3 months
  This study uses ELISA kit to measure the concentraion (pg/ml) of Leptin.
Leptin | Change from Baseline biomarkers at 4 months
  This study uses ELISA kit to measure the concentraion (pg/ml) of Leptin.
IL-1 | Change from Baseline biomarkers at 3 months
  This study uses ELISA kit to measure the concentraion (ng/ml) of interleukin-1 (IL-1).
IL-1 | Change from Baseline biomarkers at 4 months
  This study uses ELISA kit to measure the concentraion (ng/ml) of interleukin-1 (IL-1).
IL-6 | Change from Baseline biomarkers at 3 months
  This study uses ELISA kit to measure the concentraion (ng/ml) of interleukin-6 (IL-6).
IL-6 | Change from Baseline biomarkers at 4 months
  This study uses ELISA kit to measure the concentraion (ng/ml) of interleukin-6 (IL-6).
MMP-3 | Change from Baseline biomarkers at 3 months
  This study uses ELISA kit to measure the concentraion (ng/ml) of matrix metalloproteinase-3 (MMP-3).
MMP-3 | Change from Baseline biomarkers at 4 months
  This study uses ELISA kit to measure the concentraion (ng/ml) of matrix metalloproteinase-3 (MMP-3).
MMP-13 | Change from Baseline biomarkers at 3 months
  This study uses ELISA kit to measure the concentraion (pg/ml) of matrix metalloproteinase-13 (MMP-13).
MMP-13 | Change from Baseline biomarkers at 4 months
  This study uses ELISA kit to measure the concentraion (pg/ml) of matrix metalloproteinase-13 (MMP-13).
ADAMTS-4 | Change from Baseline biomarkers at 3 months
  This study uses ELISA kit to measure the concentraion (ng/ml) of a disintegrin and metalloproteinase with thrombospondin motifs-4 (ADAMTS-4).
ADAMTS-4 | Change from Baseline biomarkers at 4 months
  This study uses ELISA kit to measure the concentraion (ng/ml) of a disintegrin and metalloproteinase with thrombospondin motifs-4 (ADAMTS-4).
TG-2 | Change from Baseline biomarkers at 3 months
  This study uses ELISA kit to measure the concentraion (ng/ml) of Transglutaminase 2 (TG-2).
TG-2 | Change from Baseline biomarkers at 4 months
  This study uses ELISA kit to measure the concentraion (ng/ml) of Transglutaminase 2 (TG-2).
Metabolomics | Change from Baseline metabolomics at 3 months
  The metabolite of the drugs. This measurement used LC-MS to get the molecular weight of Chinese herbal metabolites form blood, urine and synovial fluid. This method can help to identify the active substance from the formula (TGF). Here, we cannot to know the exactly active substance that we will get.
Metabolomics | Change from Baseline metabolomics at 4 months
  The metabolite of the drugs. This measurement used LC-MS to get the molecular weight of Chinese herbal metabolites form blood, urine and synovial fluid. This method can help to identify the active substance from the formula (TGF). Here, we cannot to know the exactly active substance that we will get.
Mitochondria research--mtDNA copy number | Change from Baseline mtDNA copy number at 3 months
  mtDNA copy number
Mitochondria research--mtDNA copy number | Change from Baseline mtDNA copy number at 4 months
  mtDNA copy number
Mitochondria research--the expression of messenger ribonucleic acid in Peroxisome proliferator-activated receptor-γ coactivator-1α | Change from Baseline the expression of mRNA in PGC-1α at 3 months
  the expression of mRNA in PGC-1α by quantitative polymerase chain reaction
Mitochondria research--the expression of messenger ribonucleic acid in Peroxisome proliferator-activated receptor-γ coactivator-1α | Change from Baseline the expression of mRNA in PGC-1α at 4 months
  the expression of mRNA in PGC-1α by quantitative polymerase chain reaction
Mitochondria research--the expression of messenger ribonucleic acid in Nuclear respiratory factor 1 | Change from Baseline the expression of mRNA in NRF1 at 3 months
  the expression of mRNA in NRF1 by quantitative polymerase chain reaction
Mitochondria research--the expression of messenger ribonucleic acid in Nuclear respiratory factor 1 | Change from Baseline the expression of mRNA in NRF1 at 4 months
  the expression of mRNA in NRF1 by quantitative polymerase chain reaction
Mitochondria research--the expression of messenger ribonucleic acid in mtTFA | Change from Baseline the expression of mRNA in mtTFA at 3 months
  the expression of mRNA in mtTFA by quantitative polymerase chain reaction
Mitochondria research--the expression of messenger ribonucleic acid in mtTFA | Change from Baseline the expression of mRNA in mtTFA at 4 months
  the expression of mRNA in mtTFA by quantitative polymerase chain reaction
Mitochondria research--the expression of protein in Peroxisome proliferator-activated receptor-γ coactivator-1α | Change from Baseline the expression of protein in PGC-1α at 3 months
  the expression of protein in PGC-1α by Western blotting
Mitochondria research--the expression of protein in Peroxisome proliferator-activated receptor-γ coactivator-1α | Change from Baseline the expression of protein in PGC-1α at 4 months
  the expression of protein in PGC-1α by Western blotting
Mitochondria research--the expression of protein in Nuclear respiratory factor 1 | Change from Baseline the expression of protein in NRF1 at 3 months
  the expression of protein in NRF1 by Western blotting
Mitochondria research--the expression of protein in Nuclear respiratory factor 1 | Change from Baseline the expression of protein in NRF1 at 4 months
  the expression of protein in NRF1 by Western blotting
Mitochondria research--the expression of protein in mtTFA | Change from Baseline the expression of protein in mtTFA at 3 months
  the expression of protein in mtTFA by Western blotting
Mitochondria research--the expression of protein in mtTFA | Change from Baseline the expression of protein in mtTFA at 4 months
  the expression of protein in mtTFA by Western blotting
Mitochondria research--anti-oxidant capacity | Change from Baseline anti-oxidant capacity at 3 months
  anti-oxidant capacity by OxiSelectTM Trolox Equivalent Antioxidant Capacity (TEAC) Assay Kit (ABTS)
Mitochondria research--anti-oxidant capacity | Change from Baseline anti-oxidant capacity at 4 months
  anti-oxidant capacity by OxiSelectTM Trolox Equivalent Antioxidant Capacity (TEAC) Assay Kit (ABTS)
hsCRP | Change from Baseline CRP at 3 months
  For evaluating the status of inflammation. High-sensitivity C-reactive Protein is a protein that increases in the blood with inflammation and infection as well as following a heart attack, surgery, or trauma. Thus, it is one of several proteins that are often referred to as acute phase reactants. The high-sensitivity CRP test measures low levels of CRP in the blood to identify low levels of inflammation that are associated with risk of developing cardiovascular disease (CVD).
hsCRP | Change from Baseline CRP at 4 months
  For evaluating the status of inflammation. High-sensitivity C-reactive Protein is a protein that increases in the blood with inflammation and infection as well as following a heart attack, surgery, or trauma. Thus, it is one of several proteins that are often referred to as acute phase reactants. The high-sensitivity CRP test measures low levels of CRP in the blood to identify low levels of inflammation that are associated with risk of developing cardiovascular disease (CVD).

CONTACTS AND LOCATIONS:
Overall Officials: Hen-Hong Chang, Principal Investigator — Dean of Chinese medicine, China Medical University